CLINICAL TRIAL: NCT05951946
Title: An Open Label, 6-sequence, 3-period Study to Evaluate Drug-drug Interactions and Safety Between "BR3006-1", "BR3006-2", and "BR3006-3" in Healthy Volunteers
Brief Title: A Study to Evaluate Drug-drug Interactions and Safety Between "BR3006-1", "BR3006-2", and "BR3006-3" in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-DPMC-CT-101
Record Dates: First submitted 2023-07-06; First posted 2023-07-19 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment 1(T1) (Active Comparator): BR3006-1 + BR3006-2 administered in combination once daily for 7 days.
  Interventions: Drug: BR3006-1; Drug: BR3006-2
- Treatment 2(T2) (Active Comparator): BR3006-3 administered alone once daily for 7 days.
  Interventions: Drug: BR3006-3
- Treatment 3(T3) (Experimental): BR3006-1 + BR3006-2 + BR3006-3 administered in combination once daily for 7 days.
  Interventions: Drug: BR3006-1; Drug: BR3006-2; Drug: BR3006-3

INTERVENTIONS:
Drug: BR3006-1 — All subjects who have been fasting for at least 10 hours prior to administration will take investigational products orally with 150 mL of water at room temperature at around 8 a.m. on the administration day of each period.
  Arms: Treatment 1(T1); Treatment 3(T3)
Drug: BR3006-2 — All subjects who have been fasting for at least 10 hours prior to administration will take investigational products orally with 150 mL of water at room temperature at around 8 a.m. on the administration day of each period.
  Arms: Treatment 1(T1); Treatment 3(T3)
Drug: BR3006-3 — All subjects who have been fasting for at least 10 hours prior to administration will take investigational products orally with 150 mL of water at room temperature at around 8 a.m. on the administration day of each period.
  Arms: Treatment 2(T2); Treatment 3(T3)

SUMMARY:
The purpose of this clinical trial is to evaluate drug-drug interactions and safety between "BR3006-1", "BR3006-2", and "BR3006-3" in healthy volunteers

DETAILED DESCRIPTION:
A total of 36 subjects will be randomized into 6 sequence groups, 6 subjects per sequence group. The Investigational Products wil be according to the treatment group (A,B,C,D,E,F) assigned to each sequence group in Period 1, Period 2 and Period 3.

ELIGIBILITY:
Inclusion Criteria:

* At the time of screening test, those who weigh 55 kg or more for men and 50 kg or more for women and have body mass index (BMI) within the range of 18.5 to 30.0 kg/m2.
* Those who voluntarily decide to participate in the study after listening to and fully understanding the detailed explanation of this study and provide written consent prior to the screening procedure.

Exclusion Criteria:

* Those who have clinically significant diseases associated with the liver, kidney, gastrointestinal system, respiratory system, musculoskeletal system, endocrine system, neuropsychiatric system, blood/tumor system, cardiovascular system, severe infection, severe traumatic systemic disorder, etc.
* Those who have a medical history of gastrointestinal diseases (e.g., Crohn's disease, ulcerative disease, etc.) or gastrointestinal surgery (however, appendectomy, hernia surgery, endoscopic polyp surgery, hemorrhoids•anal fissure•anal fistula surgery are excluded) that may affect the absorption of drugs.
* Those who have participated in another clinical study within 180 days prior to the first administration date.(However, the termination criteria for participation in previous clinical trials is counted as one day after the date of the last administration)
* Those who take any prescription drugs(including herbal medicines) or any over-the-counter (OTC) drugs within 14 days prior to the first day of administration or who disagree with the prohibition about taking it from within 14 days prior to the first day of administration to the end of the study (however, if it don't affect subject's safety and study's result according to the judgment of the investigator, they may participate in the study.)
* Those who have taken a food (e.g., grapefruit juice, etc.) or health functional foods that may affect the absorption, distribution, metabolism, and excretion of the drug within 3 days prior to the first day of administration or cannot stop taking it from within 3 days prior to the first day of administration to the end of the study.
* Those who do not agree to rule out the possibility of their and their spouses' or sexual partners' pregnancy by using methods of contraception (except for hormone drugs) accepted in clinical trial from the date of the first administration of the investigational product to 7 days after the last administration or disagrees to provide their sperm or ovum

  * Methods of contraception accepted in clinical trial: Combined use of intrauterine device, vasectomy, tubal ligation, and barrier methods (male condom, female condom, cervical cap, diaphragm, sponge, etc.) or combined use of two or more barrier methods if spermicide is used
* Those who have a hereditary disorder including galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption, etc.
* Pregnant women, breast-feeding women or those positive in a pregnancy test.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-07-22 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss | Day 1 (0h), Day 5 (0h), Day 6 (0h), Day 7 (0h~14h) & Day 8 (0h), Day 9 (0h), Day 10 (0h) of each period
  Area under the concentration-time curve from time zero to time τ of BR3006-1, BR3006-2 and BR3006-3 at steady-state
Cmax,ss | Day 1 (0h), Day 5 (0h), Day 6 (0h), Day 7 (0h~14h) & Day 8 (0h), Day 9 (0h), Day 10 (0h) of each period
  Maximum concentration of drug in plasma of BR3006-1, BR3006-2 and BR3006-3 at steady-state

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Bundang Medical Center(CBMC), Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No